CLINICAL TRIAL: NCT04714008
Title: Impact of the COVID-19 Pandemic on Online Gambling in France and Sweden
Brief Title: Covid-19 and ONline GAmbling
Acronym: CONGA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0010
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Gambling; Covid19
Keywords: Gambling; Internet; Gambling tracking data; France; Sweden; Covid 19
MeSH Terms: conditions — Gambling; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active gamblers in 2019/2020: Three panels of 40 000 gamblers active in 2019 and 2020, either in France or Sweden
- Newly registered gamblers in 2019 or 2020 (France and Sweden): Six panels of 10 000 gamblers who newly registered either during the period of March-May 2019 or of March-May 2020, either in France or Sweden

SUMMARY:
The coronavirus disease 2019 (COVID-19) pandemic represents a major threat to global health. Since the beginning of the COVID-19 epidemic, all eyes have been focused on the significant somatic complications of COVID-19, but the impact on behaviors, particularly those that can lead to addictive disorders, remains little studied. A set of factors could explain a change in gambling activities, both in number of gamblers and in intensity of practices, due to the pandemic. On the one hand, the reduction or even the interruption of sporting and horse racing competitions may induce a decrease in these activities (both online and offline). Moreover, the closure of certain gambling venues and travel restrictions may also lead to a decrease of offline gambling activities in general. On the other hand, gamblers who can no longer perform their usual gambling activity could refer to available online gambling activities (poker, lotteries, casinos, etc.). Moreover, the threat of a financial crisis, the negative impact on psychological well-being (due to social isolation, stress of being infected, etc.), and increased time spent freely online, could also very largely motivate an initiation or an exacerbation of the gambling activity, especially online and in people in a situation of vulnerability. Both in France and Sweden, the closing of sports and horse race events has led to a sharp decrease in sports and horse-race betting. In both countries, the increase in other gambling types, including illegal gambling, and their potential for gambling problems is a source of concerns for public health authorities. As a consequence, more research is promptly needed in this area.

The use of gambling tracking data, widely acclaimed in recent years in research on online gambling given its ecological nature, could allow observing longitudinally changes in online gambling practices (both the raw gambling activity and risky behaviors) and in the use of responsible gambling (RG) tools due to the pandemic. Moreover, the combination of French and Swedish data will allow comparing two countries with very distinct politics regarding the pandemics, i.e. a lockdown in France in March - May 2020 and then in November - December 2020 compared to no lockdown in Sweden. Finally, gambling in women is on the rise and women display specific gambling behaviors, especially in early stages of the online gambling practice. The project will include the investigation of gender specificities both in the investigation of the impacts of the pandemic and in the comparison of French and Sweden gambling behaviors. Age, type of gambling activity and country (France / Sweden) will also be taken into account.

ELIGIBILITY:
Inclusion Criteria :

* Gamblers registered on the authorized gambling websites of France and Sweden, whatever the type of gambling activity. Those gamblers will be drawn at random from the entire active accounts datasets from the participating operators/regulatory authorities.

Exclusion Criteria :

* No exclusion criteria will be applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gamblers registered on the authorized gambling websites of France and Sweden, whatever the type of gambling activity.
Sampling Method: Probability Sample
Enrollment: 120000 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Trajectories of gambling behaviors across time before and during the pandemics | 2019-2020
  Because "gambling activity" is not directly measured as such, but rather observed as a combination of gambling indicators (e.g. money spent, type of game, numbers of gambling days, etc.), these indicators will be included as observed variables, explained by a latent (unobserved) variable, namely "gambling activity". Subgroups of gamblers with distinct impacts of the COVID-19 on their gambling activities will be identified.

SECONDARY OUTCOMES:
Typologies of gamblers based on their gambling activity and their use of RG tools outside the pandemics | 2019
  Profiles of gamblers who have similar gambling behaviors and/or use of RG tools
Gambling activity of early registered gamblers, during and outside the pandemics | 6 months after registration
  Typologies of gambling behavior trajectories across the 6 months after registration
Typologies of gamblers based on their gambling activity and their use of RG tools according to the type of gambling activity, gender, age groups and country | 2019-2020
  Profiles of gamblers who have similar gambling behaviors and/or use of RG tools, compared according to the type of gambling activity, gender, age groups and country

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Balem M, Karlsson A, Widinghoff C, Perrot B, Challet-Bouju G, Hakansson A. Gambling and COVID-19: Swedish national gambling data from a state-owned gambling sports and casino operator. J Behav Addict. 2023 Mar 30;12(1):230-241. doi: 10.1556/2006.2022.00089. Print 2023 Mar 30. PMID 36995980